CLINICAL TRIAL: NCT01668043
Title: A Phase IIa, Open-label, Multiple-Dose Trial to Investigate the Safety and Efficacy of the UB-421 in Asymptomatic HIV-1 Infected Adults
Brief Title: Study to Evaluate Safety and Efficacy of UB-421 Antibody in HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Biomedical (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Kaohsiung Veterans General Hospital. (Other); UBI Asia in Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBI Protocol A201; Protocol A201-HIV (Other: UBI Asia)
Record Dates: First submitted 2012-08-01; First posted 2012-08-17 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: HIV-1 Infection in Adults
Keywords: HIV-1; CD4; antibody; immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibody UB-421 Cohort 1 (Experimental): 10 mg/kg BW, 8 weekly doses for 8-week treatment period
  Interventions: Drug: Antibody UB-421
- Antibody UB-421 Cohort 2 (Experimental): 25 mg/kg BW, 4 biweekly doses for 8-week treatment period
  Interventions: Drug: Antibody UB-421

INTERVENTIONS:
Drug: Antibody UB-421 — UB-421 is administered by intravenous infusion

SUMMARY:
The purpose of this Phase IIa study is to determine whether the antibody (UB-421), targeting the HIV-1 receptor on the CD4 molecule of T-lymphocytes and monocytes, is safe and effective when multiple doses are administered by intravenous infusion to asymptomatic HIV-1 infected adults and to assess pharmacokinetic parameters of the antibody in blood and on cells. The neutralizing activity of UB-421 blocks HIV-1 from binding to its receptor on CD4-positive cells; thus, UB-421 functions as an immunotherapeutic intervention to prevent HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic, treatment-naive, HIV-1 seropositive
* CD4+ T cell count >350 cells/cubic millimeter
* HIV-1 viral load >5,000 copies/mL
* Other inclusion criteria apply

Exclusion Criteria:

* Active infection requiring immediate therapy (except HIV-1)
* Previous exposure to monoclonal antibody (including UB-421)
* Prior participation in any HIV vaccine trial
* Use of immunomodulating drugs or systemic chemotherapy
* Other exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of multiple intravenous infusions of two dose cohorts of UB-421 | 16-week study period
  Safety evaluations include physical examination, measurement of vital signs, clinical chemistry and hematology tests at each visit (to assess changes from normal range), incidence of adverse event (AE) and serious AE (SAE) of two dose cohorts and are followed for 16 weeks (end of study).
  Overall treatment tolerability of UB-421 for each cohort is defined as the percentage of the number of actual infusion doses divided by number of actual infusion doses plus number of missed doses of subject(s) who drops out due to drug-related AE(s); calculation follows specific formula.
To evaluate efficacy by measurement of individual maximal viral load reduction and mean maximal viral load reduction of two dose cohorts of UB-421. | 16-week study period
  Efficacy measurements include virologic responses and determination of the proportion of subjects with viral load <50 copies/mL or <200 copies/mL; viral load reduction >0.5 log10 copies/mL or >1.0 log10 copies/mL; viral rebound over 0.5 log10 increase in viral load from the nadir value during 8-week treatment period, suggesting presence of study drug resistance mutants. HIV-1 viral load is determined at each blood collection during 16-week study period.

SECONDARY OUTCOMES:
To determine pharmacokinetic parameters of two dose cohorts of UB-421. | 16-week study period
  Pharmacokinetic analyses are calculated at each visit during 8-week treatment period to determine the serum concentration before and after each infusion of UB-421 and during the 8-week follow-up period to determine the clearance of study drug in circulation.
To determine the anti-UB-421 antibody concentration in serum of two dose cohorts of UB-421 | 16-week study period
  Immunogenicity of the study drug is measured by analytical ELISA test at each visit to determine if the anti-UB-421 antibody concentration is increased above the pre-treatment baseline level.

OTHER OUTCOMES:
To determine pharmacokinetic parameters of two dose cohorts of UB-421 | 16-week study period
  Pharmacokinetic analyses are calculated at each visit during 8-week treatment period to determine the percentage of CD4+ T lymphocytes binding to the UB-421 study drug before each infusion and during the 8-week follow-up period to determine the duration of study drug bound to the CD4+ cells in circulation
To evaluate safety of multiple intravenous infusions of two dose cohorts of UB-421 | 16-week study period
  Safety evaluations include evaluation of peripheral blood mononuclear cell proliferation and expression of Th1 and Th2 cytokines in the presence of study drug before the first and last UB-421 infusions during 8-week treatment period and at the end of follow-up period.
To evaluate efficacy by measurement of individual viral load samples for appearance of drug resistance mutants in the two dose cohorts of UB-421 | 16-week period
  Efficacy measurements include virologic responses and determination of the proportion of subjects (if any) with viral load rebound during 8-week treatment period, suggesting emergence of study drug resistance mutants. Samples with viral load rebound will be characterized further to identify virus mutation(s).

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wai Wong, M.D., Principal Investigator — Taipei Veterans General Hospital (TVGH); Hung Chin Tsai, M.D., Principal Investigator — Kaohsiung Veterans General Hospital (KVGH)
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital (TVGH), Taipei, Beitou District
  - Kaohsiung Veterans General Hospital (KVGH), Kaohsiung City, Zuoying District

REFERENCES:
- [Background] Wang CY, Sawyer LS, Murthy KK, Fang X, Walfield AM, Ye J, Wang JJ, Chen PD, Li ML, Salas MT, Shen M, Gauduin MC, Boyle RW, Koup RA, Montefiori DC, Mascola JR, Koff WC, Hanson CV. Postexposure immunoprophylaxis of primary isolates by an antibody to HIV receptor complex. Proc Natl Acad Sci U S A. 1999 Aug 31;96(18):10367-72. doi: 10.1073/pnas.96.18.10367. PMID 10468614
- [Background] Lynn S and Wang CY. Designed deimmunied monoclonal antibodies for protection against HIV exposure and treatment of HIV infection. U.S. Patent No. 7,501,494. http://patft.uspto.gov/netahtml/PTO/srchnum.htm